CLINICAL TRIAL: NCT02069223
Title: Physiological Impact of Each Component of the Biliopancreatic Diversion With Duodenal Switch and Sleeve Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Johnson & Johnson (Industry); Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 21003
Record Dates: First submitted 2014-02-06; First posted 2014-02-24 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Biliopancreatic Diversion With Duodenal Switch; Gastrectomy
Keywords: Biliopancreatic Diversion with Duodenal Switch; Gastrectomy
MeSH Terms: interventions — Gastrectomy; Biliopancreatic Diversion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gastrectomy (Active Comparator): Subjects in this group will undergo a gastrectomy as their first surgery with a BPD-DS 1-year later.
  Interventions: Procedure: Gastrectomy; Procedure: BPD-DS
- BPD-DS (Active Comparator): Subjects in this group will undergo a BPD-DS as their first surgery with a gastrectomy 1-year later.
  Interventions: Procedure: Gastrectomy; Procedure: BPD-DS
- Gastrectomy+BPD-DS (Active Comparator): Subjects in this group will undergo a gastrectomy AND a BPD-DS concomitantly. They will then be closely monitored for the remainder of the study.
  Interventions: Procedure: Gastrectomy; Procedure: BPD-DS

INTERVENTIONS:
Procedure: Gastrectomy
Procedure: BPD-DS
  Other Names: Biliopancreatic Diversion with Duodenal Switch

SUMMARY:
Bariatric surgery procedures promote weight loss by limiting the amount of food consumed through reduction of the size of the stomach and by decreasing absorption of nutrients through reorganizing or bypassing portions of the small intestine. Among the procedures used to induce weight loss, sleeve gastrectomy (SG) was initially developed in the early 90's as the restrictive component of a biliopancreatic diversion with duodenal switch (BPD-DS). It was then offered by laparoscopy as a staged-approach in order to reduce peri-operative complications in high-risk patients. The second step of the surgery (i.e. the duodenal switch) was planned when sufficient weight loss had been obtained. However, it was observed that some patients experienced appreciable weight loss with the SG alone, and did not require a second-stage surgery, thus avoiding the side-effects of a malabsorptive surgery. This led to the surge in popularity of SG as a stand-alone operation, because of its relative technical simplicity, feasibility, and good outcomes. Multiple mechanisms have been postulated to induce metabolic recovery and weight loss following surgery. The independent effects of each component of the BPD-DS with SG have never been investigated in humans within a well-controlled study design. The general objective of the present project is to assess the impact of each component of the BPD-DS and SG, either combined of separated, on physiological variables potentially responsible for metabolic recovery. Patients will be randomized to undergo one of three surgical sequences: 1) SG followed by BPD-DS one year later; 2) BPD-DS followed by SG one year later; or 3) SG and BPD-DS within a single operation. A series of tests will be performed at baseline, at 1 year, and 2 years after the initial surgery. We propose two Specific Aims to asses 1) the impact of each surgical component on the hormonal determinants of metabolic recovery; and 2) the impact of weight loss responses on subcutaneous and visceral adipose tissue function improvements. This project will help better understand the mechanisms underlying metabolic recovery following weight loss surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women between 18-60 years old;
* BMI ≥ 45 à ≤ 55 kg/m2;
* Subjects capable of understanding and being able to sign a consent form;
* Subjects capable of following the protocol directives, including the proposed visits (timeline);
* Subjects living within a reasonable distance from the hospital and capable of being present at all required visits.

Exclusion Criteria:

* Pregnant women or women who plan on becoming pregnant during the study, or women in fertile age range who refuse proper contraceptive methods during the study. (Must have negative pregnancy test at the moment of enrollment and use medically acceptable contraception which include: oral contraceptives, injectable or implantable contraceptives, intrauterine devices or double-barrier method ie. condoms and diaphragm);
* Diabetics
* Subjects with HbA1c ≥ 6,5 % or fasting Glucose ≥7mmol/l or non-fasting Glucose ≥11mmol/l;
* Previous oesophagal, gastric or bariatric surgery;
* Irritable bowel syndrome, unexplained intermittent vomiting, severe abdominal pain, diarrhea or chronic constipation;
* History of duodenal or gastric ulcers;
* Pre-operative hypoalbuminuria (<35g/l);
* History of renal disease, hepatic disease (cirrhosis) or severe cardiac or pulmonary disease;
* Corticosteroid intake in the previous month;
* Presence of psychiatric problems or behavioral issues that could limit subject's capacity at understanding the procedure and to conform to medical/surgical recommendations;
* History of drug use or alcoholism in previous 12 months before study;
* History of inflammatory diseases of the gastro-intestinal tract (Esophagitis, varices, gastric or duodenal ulcers, Crohn's disease, congenital or acquired anomalies of the digestive tract).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Measure the changes in Satiety Levels and the changes in Incretin Levels | Baseline, 12, 24 months
  * Satiety determination via questionnaires
  * Incretin levels
Measure the changes of adipose tissue cells sizes and macrophage infiltration | Baseline, 12 months
  * Adipose Tissue cell sizing
  * Adipose Tissue macrophage infiltration via histology

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUCPQ, Québec, Quebec, Canada